CLINICAL TRIAL: NCT07258576
Title: The Effect of Menstrual Cycle Phase and Oral Contraceptive Use on Muscle Protein Metabolism Post-Resistance Training
Brief Title: Menstrual Cycle vs. Oral Contraceptives: Effects on Muscle Protein Metabolism After Resistance Exercise
Acronym: MCOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MCOC - REB00048059
Record Dates: First submitted 2025-08-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Female Sex Hormones; Menstrual Cycle; Oral Contraceptives; Protein Metabolism
Keywords: Protein Metabolism; Female Sex Hormones; Menstrual Cycle; Oral Contraceptives; Resistance Exercise; Weightlifting; Indicator Amino Acid Oxidation; Stable Isotope Tracer

STUDY DESIGN:
Intervention Model Description: Between-Subject Crossover Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mid-Luteal Phase (Other): 5-9 days post-ovulation
  Interventions: Dietary Supplement: Protein Beverage; Dietary Supplement: Stable Isotope Tracer [D5]phenylalanine; Dietary Supplement: Stable Isotope Tracer [13C]phenylalanine
- Early Follicular Phase (Other): Days 2-6 post-menses onset
  Interventions: Dietary Supplement: Protein Beverage; Dietary Supplement: Stable Isotope Tracer [D5]phenylalanine; Dietary Supplement: Stable Isotope Tracer [13C]phenylalanine
- Active Pill Phase (Other): Days 10-20 of active pill
  Interventions: Dietary Supplement: Protein Beverage; Dietary Supplement: Stable Isotope Tracer [D5]phenylalanine; Dietary Supplement: Stable Isotope Tracer [13C]phenylalanine
- Placebo Pill Phase (Other): At least 48h after last active pill is taken
  Interventions: Dietary Supplement: Protein Beverage; Dietary Supplement: Stable Isotope Tracer [D5]phenylalanine; Dietary Supplement: Stable Isotope Tracer [13C]phenylalanine

INTERVENTIONS:
Dietary Supplement: Protein Beverage — Participants will consume 16 half-hourly (8 hours) isoenergetic, isonitrogenous beverages containing 1.2 g/kg/d protein.
Dietary Supplement: Stable Isotope Tracer [D5]phenylalanine — Protein beverages will be enriched with the stable isotope [D5]phenylalanine. The use of [D5]phenylalanine will allow for determination of muscle protein synthesis.
Dietary Supplement: Stable Isotope Tracer [13C]phenylalanine — Protein beverages will be enriched with the stable isotope tracer [13C]phenylalanine. The use of [13C]phenylalanine will allow for the determination of the fate of amino acids in the body (incorporation into body protein or oxidation) which can be used to determine protein requirements.

SUMMARY:
The muscles of the body are constantly breaking down old proteins and building new ones. These two processes, protein breakdown and protein synthesis, together are known as protein turnover. Protein turnover is essential for maintaining healthy muscle.

Despite its importance, females have historically been underrepresented in protein metabolism research. A long-standing assumption has been that fluctuations in female sex hormones such as estrogen and progesterone, whether across the natural menstrual cycle or in individuals using oral contraceptives (OCs), make metabolism and training responses too variable to study. Because of this, many researchers have excluded female participants for logistical reasons.

Resistance exercise, such as weightlifting, is the most effective way to increase muscle size and strength. Each resistance-training session triggers muscle protein synthesis (MPS), the process by which new muscle proteins are built. Consuming dietary protein or individual amino acids further increases the rate at which new proteins are formed. Over time, higher rates of protein synthesis support muscle growth and the maintenance of other lean tissues in the body.

The purpose of this study is to examine how menstrual cycle phases and OC use influence the synthesis of proteins in both muscle tissue and the rest of the body. Improving scientific understanding in this area will support more effective, evidence-based training and nutrition recommendations for females.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* BMI between 18.5-29.9 kg/m2 (non-obese)
* Recreationally active (resistance train minimum twice a week)
* Using monophasic or triphasic oral contraceptives for >1 year (for oral contraceptive users)
* Have regular menstrual cycles (21-35 days) for the past 3 months and discontinued any hormonal contraceptive use for at least 6 months (non-oral contraceptive users)
* Must meet a progesterone sufficiency test (non-oral contraceptive users)

Exclusion Criteria:

* Mid-luteal progesterone levels <16umol
* Chronic disease diagnosis (cardiovascular, thyroid, diabetes)
* Current or recent remission of cancer
* Regular use of non-steroidal anti-inflammatory drugs (NSAIDs; except low-dose aspirin), anticoagulants
* Use of prescription drugs that would impact muscle protein synthesis, e.g. Statins, Lithium, ADHD medication.
* Insertion of intrauterine device (IUD) - exception: copper
* Use of emergency contraception in the last 3 months (e.g. Plan B)
* Severe food allergies (e.g. soy, nuts)
* Smoking, use of performance enhancing drugs (growth hormones, testosterone)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-females with regular menses or using oral contraceptives.
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis (MPS) | 8 hours
  Muscle protein synthesis (MPS) will be assessed during an 8-hour post-exercise and feeding period using a stable isotope tracer, L-[ring-D5]phenylalanine ([D5]Phe). The incorporation of the [D5]Phe tracer into myofibrillar muscle proteins, collected from muscle biopsies (pre-exercise and post-8h feeding), will be analyzed using liquid chromatography-tandem mass spectrometry (LC-MS/MS) to determine the fractional synthesis rate (FSR) of muscle proteins. This will help us understand how menstrual cycle phases and oral contraceptive use influence MPS, providing insight into optimizing protein intake and training adaptations in female athletes.

SECONDARY OUTCOMES:
Whole Body Protein Synthesis (WBPS) | 4 hours
  Whole body protein synthesis (WBPS) will be measured over a 4-hour period using the Indicator Amino Acid Oxidation (IAAO) methodology. Participants will consume a stable isotope tracer, L-[1-13C]phenylalanine ([13C]Phe), and breath samples will be collected every 30 minutes during the final 4 hours of the metabolic trial. The enrichment of 13CO₂ in breath samples will be analyzed to determine phenylalanine oxidation rates, providing an estimate of whole-body protein turnover and dietary protein utilization. This will allow us to assess whether hormonal fluctuations influence protein metabolism and nutritional requirements in female athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Center for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided